CLINICAL TRIAL: NCT06712758
Title: Low Intraocular Pressure Cataract Surgery With Zeiss Quatera in Glaucoma Patients. Prospective, Investigator Initiated and Observational Case Series
Brief Title: Low Intraocular Pressure Cataract Surgery With Zeiss Quatera in Glaucoma Patients
Status: Recruiting | Type: Observational
Sponsor: Visionair Oogzorg (Other)
Responsible Party: Principal Investigator, Koen Willekens, Professor Doctor, Visionair Oogzorg
Other Study IDs: Quatera
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Cataract; Glaucoma
Keywords: intra ocular pressure; cataract; Quatera; glaucoma
MeSH Terms: conditions — Cataract; Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Glaucoma patients in need of cataract surgery: Cataract surgery

SUMMARY:
You were selected to participate in this observational study because you suffer from glaucoma and cataracts. For the cataract you will have cataract surgery. This study will not affect your treatment, it will only collect data on what is performed before, during and after the procedure.

The aim of this data collection is to demonstrate the safety of a new generation of cataract surgical devices in patients who also suffer from glaucoma. They are glaucoma patients who have an increased sensitivity to eye pressure increases both during and after surgery. The new surgical device makes it possible to safely perform cataract surgery under low pressures. This could, at least theoretically, provide an advantage for patients who also suffer from glaucoma.

DETAILED DESCRIPTION:
Cataract surgery is a highly standardized procedure. However a new phacoemulsification system "Quatera 700" has been developed by Carl Zeiss Meditec. The system has a unique patented QUATTRO Pump that directly controls infusion and aspiration and enables a synchronous change in both. It has four membranes, which directly regulate infusion and aspiration and maintain a pre-set intraocular pressure (IOP), resulting in a stable anterior chamber during the surgery. The membranes are activated by pneumatic pressure regulated by sensors that measure infusion and aspiration flows which allows the system to determine and compensate for incisional leakage as well. This innovative pump system allows surgeons to significantly decrease the intra-ocular pressure during cataract surgery. In respect to competitive devices on the market, the Quatera system is able to operate with pressure four times lower than average. Especially in glaucoma patients (patients suffering from optic nerve head damage due to elevated intraocular pressures), performing surgery with lower intra-ocular pressures would help in avoiding extra nerve fiber layer damage and overall safety of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with glaucoma that are diagnosed with age-related cataract

Exclusion Criteria:

* Unwilling to sign informed consent
* Functionally monophtalmic patient
* Endothelial dystrophy
* Active uveitis
* Known corticosteroid responder
* Presence of uncontrolled systemic disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from Dr. Koen Willekens at Visionair Oogzorg.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Complication rate during cataract surgery | Month 1
  Complication rate during cataract surgery

SECONDARY OUTCOMES:
Best corrected visual acuity | Month 1
  Best corrected visual acuity will be determined and recorded at the preoperative, day 1, week
  1 and month 1 visit.
Intraocular pressure | 1 month
  The intraocular pressure will be measured at the preoperative, day 1, week 1 and month 1 visit. Ocular hypertension will reported.
Retinal nerve fiber layer thickness | 1 year
  Optical Coherence Tomography will be performed at the preoperative and month 1 visit. Any abnormalities will be described.
Visual field mean deviation | Month 1
  The visual field examination will be performed at the preoperative and month 1 visit. Any abnormalities will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Willekens, Principal Investigator — Visionair Oogzorg
Locations (1):
- Visionair Oogzorg, Geel, Belgium

IPD SHARING:
Plan to Share IPD: Undecided